CLINICAL TRIAL: NCT03893669
Title: Randomized, Double-blinded, Controlled, Phase I Trial to Assess Safety, Tolerability and Immunogenicity of 'NBP607(Trivalent Inactivated Cell-Culture Influenza Vaccine)' Compared to Egg-based Influenza Vaccine in Healthy Adult
Brief Title: Safety, Tolerability and Immunogenicity of an Trivalent Inactivated Cell-Culture Influenza Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NBP607_Flu_I_2012
Record Dates: First submitted 2012-12-12; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2012-10

CONDITIONS: Prevention of Influenza

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): NBP607 0.5ml
  Interventions: Biological: NBP607
- Group 2 (Active Comparator): Agrippal 0.5ml
  Interventions: Biological: Agrippal

INTERVENTIONS:
Biological: NBP607 — 1 dose, 0.5ml, Intramuscular (IM) injection
  Arms: Group 1
Biological: Agrippal — 1 dose, 0.5ml, Intramuscular (IM) injection
  Arms: Group 2

SUMMARY:
A randomized, double-blinded, controlled, Phase I clinical trial to assess the safety, tolerability and immunogenicity of 'NBP607(trivalent inactivated cell-culture influenza vaccine)' compared to egg-based influenza vaccine in healthy adult volunteers

DETAILED DESCRIPTION:
1. Assessment of Safety
2. Assessment of Immunogenicity
3. Estimated Enrollment: 100

ELIGIBILITY:
Inclusion Criteria:

1. 20 to <60 years of age
2. able and willing to give written informed consent prior to study entry
3. if female, at least 2 years after post- menopausal and negative result of urine-human chorionic gonadotropin (HCG) test at screening

Exclusion Criteria:

1. hypersensitivity to any component of the study medication or chemically related substances, such as allergy to eggs or egg products
2. Immunodeficiency disease
3. history of hypersensitivity when vaccination, such as Guillain-Barre syndrome
4. thrombocytopenia or Coagulation disorders
5. experienced fever (>37.5°C) within the past 24 hours or any acute respiratory infection
6. receipt of Immunosuppressants or Immunomodulators within the past 3 months
7. receipt of blood products or immunoglobulin within the past 3 months
8. received influenza vaccine within the past 6 months
9. received another vaccine within the past 1 month or plans vaccination within 1 months following the study vaccination
10. participation on another clinical trial within 1 month prior to the study vaccination
11. history of blood donation within 1 week prior to the study vaccination for plan of blood donation within 7 days following the study vaccination
12. any chronic diseases that interfere with the clinical trial or Malignant tumors
13. pregnant or breastfeeding
14. any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives or might interfere with the safety of the study subject.

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2012-09; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Incidence rate of solicited local adverse events (AEs) | Within 21 days after vaccination
  All AEs were classified and analyzed according to its severity and causality. The number and percentage of subjects with AEs were analyzed. Incidence rate, 95% confidence interval as well as number of occurrences were calculated.
Incidence rate of solicited systemic AEs | Within 21 days after vaccination
  All AEs were classified and analyzed according to its severity and causality. The number and percentage of subjects with AEs were analyzed. Incidence rate, 95% confidence interval as well as number of occurrences were calculated.
Incidence rate of unsolicited AEs | Within 21 days after vaccination
  All AEs were classified and analyzed according to its severity and causality. The number and percentage of subjects with AEs were analyzed. Incidence rate, 95% confidence interval as well as number of occurrences were calculated.
Pulse rate at each visit | 0-14 days prior to vaccination/day of vaccination/3-7 days after vaccination/21-28 days after vaccination
  Comparisons within each group between pre-/post- vaccination were summarized and presented.
Blood pressure(systolic/diastolic) at each visit | 0-14 days prior to vaccination/day of vaccination/3-7 days after vaccination/21-28 days after vaccination
  Comparisons within each group between pre-/post- vaccination were summarized and presented.
Body temperature at each visit | 0-14 days prior to vaccination/day of vaccination/3-7 days after vaccination/21-28 days after vaccination
  Comparisons within each group between pre-/post- vaccination were summarized and presented.
Rate of normal/abnormal results in Electrocardiogram (ECG) (ventricular rate, PR interval, QRS, QT, and QTc) collected during screening visit and close-out visit | Screening visit(0-14 days prior to vaccination)/close-out visit(21-28 days after vaccination)
  Comparisons within each group between pre-/post- vaccination were summarized and presented.
Rate of normal/abnormal results in physical examination at each visit | 0-14 days prior to vaccination/day of vaccination/3-7 days after vaccination/21-28 days after vaccination
  Comparisons within each group between pre-/post- vaccination were summarized and presented.
Rate of normal/abnormal results in clinical laboratory tests(Platelet, Cl, etc.) during screening visit and close-out visit | Screening visit(0-14 days prior to vaccination)/close-out visit(21-28 days after vaccination)
  Comparisons within each group between pre-/post- vaccination were summarized and presented.

SECONDARY OUTCOMES:
Seroconversion rate measured by pre-/post-vaccination Haemagglutination Inhibition (HI) titer[Immunogenicity] | 21-28 days after vaccination
  The proportion of subjects achieving one of the following conditions; i)If the pre-vaccination HI titer were <1:10, subjects achieving an HI titer ≥1:40 after vaccination ii)If the pre-vaccination HI titers were ≥1:10, subjects with a minimum 4-fold rise in HI titer
Geometric Mean Ratio (GMR) measured by pre-/post-vaccination HI titer[Immunogenicity] | 21-28 days after vaccination
  The mean increase in geometric mean HI titer
Seroprotection rate measured by post-vaccination HI titer[Immunogenicity] | 21-28 days after vaccination
  The proportion of subjects with post-vaccination HI titers of ≥1:40

CONTACTS AND LOCATIONS:
Overall Officials: Woo Joo Kim, Ph.D., Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, Guro-gu, South Korea